CLINICAL TRIAL: NCT04782154
Title: Paceport Swan-Ganz Data Collection Study
Status: Completed | Type: Observational
Sponsor: Montreal Heart Institute (Other)
Collaborators: Edwards Lifesciences (Industry)
Responsible Party: Principal Investigator, Andre Denault, MD, PhD, FRCPC, ABIM-CC, Montreal Heart Institute
Other Study IDs: 2018-20
Record Dates: First submitted 2021-03-01; First posted 2021-03-04 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Right Ventricular Dysfunction; Right Heart Failure; Congestive Heart Failure
Keywords: Right Ventricular Pressure Waveform
MeSH Terms: conditions — Ventricular Dysfunction, Right; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
RV dysfunction has been associated with increased mortality in the ICU and cardiac surgical patients. Thus, early identification of RV dysfunction at less severe stages will allow for earlier intervention and potentially better patient outcomes. However, so far, no studies have reported prospectively the prevalence of abnormal RV pressure waveform during cardiac surgery and in the ICU. Our primary hypothesis is that the prevalence of abnormal RV pressure waveform occurs in more than 50% of cardiac surgical patients throughout their hospitalization. Those patients with abnormal RV pressure waveform will be more prone to post-operative complications related to RV dysfunction and failure in the OR and ICU.

DETAILED DESCRIPTION:
The pulmonary artery catheter (PAC) consists of an intravenous device placed in the pulmonary artery to measure cardiac output, pulmonary artery pressures (Richard C, 2011) as well as cardiac filling pressures. Since its initial presentation by Swan in 1970 (H J Swan, 1970), several modifications were made on the initial catheter now allowing continuous assessment of cardiac output, continuous monitoring of stroke volume (SV), systemic vascular resistance (SVR) and mixed venous saturation (SvO2) (Arora, 2014) (H J Swan, 1970) (Richard C, 2011). We intend to enhance current Swan-Ganz catheters with clinical decision support tools to early identify hemodynamically unstable states that can lead to further deterioration of the patient's health state.

Right ventricular (RV) dysfunction is mostly associated to a decrease in contractility, right ventricular pressure overload or right ventricular volume overload (François Haddad, 2008). RV dysfunction can occur in several clinical scenarios in the intensive care unit (ICU) and operating room (OR): pulmonary embolism, acute respiratory distress syndrome (ARDS), septic shock, RV infarction, and in pulmonary hypertensive patients undergoing cardiac surgery (François Haddad, 2008). RV dysfunction has been associated with increased mortality in the ICU and cardiac surgical patients (André Y. Denault, 2006) (Denault AY B. J.-S., 2016). Thus, early identification of RV dysfunction at less severe stages will allow for earlier intervention and potentially better patient outcomes. Unfortunately, identifying which patients will develop RV dysfunction and then progress towards RV failure have proven difficult. One of the reasons for delaying the diagnosis of RV dysfunction could be the lack of uniform definition, especially in the perioperative period. Echocardiographic definitions of RV dysfunction have been described in previous studies: RV fractional area change (RVFAC) < 35 %, tricuspid annular plane systolic excursion (TAPSE) < 16 mm, tissue Doppler S wave velocity <10 cm/s, RV ejection fraction (RVEF) <45% and RV dilation have been related to RV dysfunction (Rudski LG, 2010). However, these echocardiographic indices cannot be continuously monitored and are insufficient in describing RV function. The diagnosis of fulminant RV failure is more easily recognized as a combination of echocardiographic measures, compromised hemodynamic measures and clinical presentation (Raymond M, 2019) (François Haddad, 2008) (Haddad F, 2009). RV dysfunction is inevitably associated with absolute or relative pulmonary hypertension because of the anatomic and physiological connection between the RV and pulmonary vascular system (Naeije R, 2014) (François Haddad, 2008). The gold standard for measuring pulmonary pressure is still the pulmonary artery catheter. However, RV output can initially be preserved despite of pulmonary hypertension (Denault AY C. M., 2006). It is therefore mandatory that early, objective, continuous, easily obtainable and subclinical indices of RV dysfunction are found and validated to initiate early treatment of this disease.

Since 2002, Dr Denault's group at Montreal Heart Institute has been using continuous RV pressure waveform monitoring initially for the diagnosis of RV outflow tract obstruction (Denault A, 2014) and then for RV diastolic dysfunction evaluation (St-Pierre P, 2014) (Myriam Amsallem, 2016). Preliminary data based on a retrospective study on 259 patients found that 110 (42.5%) patients had abnormal RV gradients before cardiopulmonary bypass (CPB).Abnormal RV diastolic pressure gradient was associated with higher EuroSCORE II (2.29 [1.10-4.78] vs. 1.62 [1.10-3.04], p=0.041), higher incidence of RV diastolic dysfunction using echocardiography (45 % vs. 29 %, p=0.038), higher body mass index (BMI) (27.0 [24.9-30.5] vs. 28.9 [25.5-32.5], p=0.022), pulmonary hypertension (mean pulmonary artery pressure (MPAP) > 25 mmHg) (37 % vs. 48 %, p=0.005) and lower pulmonary artery pulsatility index (PAPi) (1.59 [1.19-2.09] vs. 1.18 [0.92-1.54], p<0.0001). Patients with abnormal RV gradient had more frequent difficult separation from CPB (32 % vs. 19 %, p=0.033) and more often received inhaled pulmonary vasodilator treatment before CPB (50 % vs. 74 %, p<0.001). However, this was retrospective and limited to the pre-CPB period.

In 2017, in a review article on RV failure in the ICU (Hrymak C, 2017), RV pressure waveform monitoring using the paceport of the pulmonary artery catheter was recommended as a simple method of monitoring RV function (Rubenfeld GD, 1999). However, no studies have reported prospectively the prevalence of abnormal RV pressure waveform during cardiac surgery and in the ICU.

ELIGIBILITY:
Inclusion Criteria:

* Be ≥ 18 years of age
* Participate in the Informed Consent process and sign/date the approved informed consent forms
* Projected to receive Swan-Ganz catheter as part of procedure/standard of care with intermittent cardiac output and mixed venous oxygen saturation (SvO2) measures

Exclusion Criteria:

* Refuse to sign consent
* Have left bundle branch block
* Have recurrent sepsis
* Have hypercoagulopathy
* Allergic to FORE-SIGHT Elite sensor adhesive
* Latex allergy due to presence of latex in the Swan-Ganz catheter balloon.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects ≥ 18 years of age, with planned surgery or liver transplantation, projected to receive Swan-Ganz as part of the procedure/standard of care with intermittent cardiac output measures will be screened for inclusion into the Study. Only subjects meeting all inclusion criteria will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2021-08-09 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Proportion of abnormal diastolic RV waveforms before CPB, after CPB and in the ICU | From thermodilution catheter insertion until 2 hours after ICU arrival
  Abnormal RV pressure waveform will be defined as a difference between the RV end-diastolic minus the early-diastolic pressure > 4 mmHg and a RVdP/dt < 400 mmHg.

SECONDARY OUTCOMES:
Proportion of patients with difficult and complex separation from cardiopulmonary bypass at the end of cardiac surgery | From the discontinuation of cardiopulmonary bypass until ICU arrival after surgery, assessed up to 4 hours
  Difficult separation from cardiopulmonary bypass: instability requiring at least two different types of pharmacological agents (i.e., inotropes ± vasopressors ± inhaled agents) Complex separation from cardiopulmonary bypass: Hemodynamic instability requiring return on cardiopulmonary bypass or addition of mechanical support (intra-aortic balloon pump or extra-corporeal membrane oxygenator)
Cumulative time of Persistent Organ Dysfunction or Death (TPOD) during the first 28 days after cardiac surgery | Up to 28 days or until hospital discharge
  TPOD is a continuous variable representative of the burden of care and morbidity during the first 28 days following cardiac surgery and was chosen to circumvent issues arising for using other clinical endpoint such as ICU length of stay
Incidence of deaths during hospitalisation | Up to 28 days or until hospital discharge
  Death from any cause
Incidence of acute kidney injury (AKI) | Up to 28 days or until hospital discharge
  Acute kidney injury (AKI) according to KDIGO serum creatinine criteria: Stage 1: ≥50% or 27 umol/L increases in serum creatinine, Stage 2: ≥100% increase in serum creatinine, Stage 3 ≥200% increase in serum creatinine or an increase to a level of ≥254 umol/L or dialysis initiation.
Incidence of major bleeding | Up to 28 days or until hospital discharge
  Major bleeding is defined by the Bleeding Academic Research Consortium (BARC) as one of the following: • Perioperative intracranial bleeding within 48h • Reoperation after closure of sternotomy for the purpose of controlling bleeding • Transfusion of ≥5 units of whole blood of packed red blood cells within a 48 hours period • Chest tube output ≥2L within a 24 hours period
Incidence of surgical reintervention for any reasons | Up to 28 days or until hospital discharge
  Re-operation after the initial surgery for any cause
Incidence of deep sternal wound infection or mediastinitis | Up to 28 days or until hospital discharge
  Diagnosis of a deep incisional surgical site infection or mediastinitis by a surgeon or attending physician
Incidence of delirium | Up to 28 days or until hospital discharge
  Delirium is defined as an intensive care delirium screening checklist (ICDSC) score(18) of ≥4 in the week following surgery or positive result for the Confusion Assessment Method for the ICU (CAM-ICU).
Incidence of stroke | Up to 28 days or until hospital discharge
  Central neurologic deficit persisting longer than 72 hours
Total duration of ICU stay in hours | Up to 28 days or until hospital discharg
  Number of hours passed in the ICU
Duration of vasopressor requirements (in hours) | Up to 28 days or until hospital discharge
  Vasopressors include norepinephrine, epinephrine, dobutamine, vasopressin, phenylephrine, milrinone, isoproterenol and dopamine
Up to 28 days or until hospital discharge | Up to 28 days or until hospital discharge
  Number of days hospitalized from the day of surgery to discharge
Duration of mechanical ventilation (in hours) | Up to 28 days or until hospital discharge
  A duration of >24 hours will be considered prolonged ventilation requirements.
Incidence of major morbidity or mortality | Up to 28 days or until hospital discharge
  Including death, prolonged ventilation, stroke, renal failure (Stage ≥2), deep sternal wound infection and reoperation for any reason.
Right ventricular ejection fraction | From arrival to the operating room until 2 hours after ICU arrival
  Assessed by the American Society of Echocardiography guidelines
Right ventricular fractional area change | From arrival to the operating room until 2 hours after ICU arrival
  Assessed by the American Society of Echocardiography guidelines
Right ventricular strain | From arrival to the operating room until 2 hours after ICU arrival
  Assessed by the American Society of Echocardiography guidelines
Tricuspid annular plane systolic excursion | From arrival to the operating room until 2 hours after ICU arrival
  Assessed by the American Society of Echocardiography guidelines
Right ventricular performance index | From arrival to the operating room until 2 hours after ICU arrival
  Assessed by the American Society of Echocardiography guidelines
Portal flow pulsatility fraction | From arrival to the operating room until 2 hours after ICU arrival
  Portal flow pulsatility fraction
Right ventricular stroke work index | From arrival to the operating room until 2 hours after ICU arrival
  0.0136x Stroke volume index x (Mean pulmonary artery pressure-mean right atrial pressure)
Relative pulmonary pressure | From arrival to the operating room until 2 hours after ICU arrival
  The ratio of the mean systemic arterial pressure divided by the mean pulmonary artery pressure
Right ventricular function index | From arrival to the operating room until 2 hours after ICU arrival
  Defined as (isovolumic contraction time + isovolumic relaxation time)/RV ejection time
Pulmonary artery pulsatility index (PAPi) | From arrival to the operating room until 2 hours after ICU arrival
  Defined as (systolic pulmonary artery pressure - diastolic pulmonary artery pressure)/central venous pressure
Compliance of the pulmonary artery (CPA) | From arrival to the operating room until 2 hours after ICU arrival
  Stroke volume divided by the pulmonary artery pulse pressure (systolic minus the diastolic pulmonary artery pressure)
Pulsatility of femoral venous flow | From arrival to the operating room until 2 hours after ICU arrival
  Velocity variations of blood flow in the femoral vein during the cardiac cycle
Right ventricular outflow tract obstruction | From arrival to the operating room until 2 hours after ICU arrival
  Right Ventricular Systolic pressure minus Pulmonary Artery Systolic pressure ≤ 6 mmHg.

CONTACTS AND LOCATIONS:
Overall Officials: Andre Y Denault, MD,PhD, Principal Investigator — Montreal Heart Institute
Locations (1):
- Montreal Heart Institute, Montreal, Quebec, Canada

REFERENCES:
- [Background] Denault AY, Couture P, Buithieu J, Haddad F, Carrier M, Babin D, Levesque S, Tardif JC. Left and right ventricular diastolic dysfunction as predictors of difficult separation from cardiopulmonary bypass. Can J Anaesth. 2006 Oct;53(10):1020-9. doi: 10.1007/BF03022532. PMID 16987858
- [Background] Mehta Y, Arora D. Newer methods of cardiac output monitoring. World J Cardiol. 2014 Sep 26;6(9):1022-9. doi: 10.4330/wjc.v6.i9.1022. PMID 25276302
- [Background] Denault A, Lamarche Y, Rochon A, Cogan J, Liszkowski M, Lebon JS, Ayoub C, Taillefer J, Blain R, Viens C, Couture P, Deschamps A. Innovative approaches in the perioperative care of the cardiac surgical patient in the operating room and intensive care unit. Can J Cardiol. 2014 Dec;30(12 Suppl):S459-77. doi: 10.1016/j.cjca.2014.09.029. Epub 2014 Oct 5. PMID 25432139
- [Background] Denault AY, Bussieres JS, Arellano R, Finegan B, Gavra P, Haddad F, Nguyen AQN, Varin F, Fortier A, Levesque S, Shi Y, Elmi-Sarabi M, Tardif JC, Perrault LP, Lambert J. A multicentre randomized-controlled trial of inhaled milrinone in high-risk cardiac surgical patients. Can J Anaesth. 2016 Oct;63(10):1140-1153. doi: 10.1007/s12630-016-0709-8. Epub 2016 Jul 28. PMID 27470232
- [Background] Denault AY, Chaput M, Couture P, Hebert Y, Haddad F, Tardif JC. Dynamic right ventricular outflow tract obstruction in cardiac surgery. J Thorac Cardiovasc Surg. 2006 Jul;132(1):43-9. doi: 10.1016/j.jtcvs.2006.03.014. PMID 16798301
- [Background] Haddad F, Hunt SA, Rosenthal DN, Murphy DJ. Right ventricular function in cardiovascular disease, part I: Anatomy, physiology, aging, and functional assessment of the right ventricle. Circulation. 2008 Mar 18;117(11):1436-48. doi: 10.1161/CIRCULATIONAHA.107.653576. No abstract available. PMID 18347220
- [Background] Swan HJ, Ganz W, Forrester J, Marcus H, Diamond G, Chonette D. Catheterization of the heart in man with use of a flow-directed balloon-tipped catheter. N Engl J Med. 1970 Aug 27;283(9):447-51. doi: 10.1056/NEJM197008272830902. No abstract available. PMID 5434111
- [Background] Haddad F, Couture P, Tousignant C, Denault AY. The right ventricle in cardiac surgery, a perioperative perspective: II. Pathophysiology, clinical importance, and management. Anesth Analg. 2009 Feb;108(2):422-33. doi: 10.1213/ane.0b013e31818d8b92. PMID 19151265
- [Background] Hrymak C, Strumpher J, Jacobsohn E. Acute Right Ventricle Failure in the Intensive Care Unit: Assessment and Management. Can J Cardiol. 2017 Jan;33(1):61-71. doi: 10.1016/j.cjca.2016.10.030. Epub 2016 Nov 11. PMID 28024557
- [Background] Amsallem M, Kuznetsova T, Hanneman K, Denault A, Haddad F. Right heart imaging in patients with heart failure: a tale of two ventricles. Curr Opin Cardiol. 2016 Sep;31(5):469-82. doi: 10.1097/HCO.0000000000000315. PMID 27467173
- [Background] Naeije R, Manes A. The right ventricle in pulmonary arterial hypertension. Eur Respir Rev. 2014 Dec;23(134):476-87. doi: 10.1183/09059180.00007414. PMID 25445946
- [Background] Raymond M, Gronlykke L, Couture EJ, Desjardins G, Cogan J, Cloutier J, Lamarche Y, L'Allier PL, Ravn HB, Couture P, Deschamps A, Chamberland ME, Ayoub C, Lebon JS, Julien M, Taillefer J, Rochon A, Denault AY. Perioperative Right Ventricular Pressure Monitoring in Cardiac Surgery. J Cardiothorac Vasc Anesth. 2019 Apr;33(4):1090-1104. doi: 10.1053/j.jvca.2018.08.198. Epub 2018 Aug 25. PMID 30269893
- [Background] Richard C, Monnet X, Teboul JL. Pulmonary artery catheter monitoring in 2011. Curr Opin Crit Care. 2011 Jun;17(3):296-302. doi: 10.1097/MCC.0b013e3283466b85. PMID 21499096
- [Background] Rubenfeld GD, Angus DC, Pinsky MR, Curtis JR, Connors AF Jr, Bernard GR. Outcomes research in critical care: results of the American Thoracic Society Critical Care Assembly Workshop on Outcomes Research. The Members of the Outcomes Research Workshop. Am J Respir Crit Care Med. 1999 Jul;160(1):358-67. doi: 10.1164/ajrccm.160.1.9807118. No abstract available. PMID 10390426
- [Background] Rudski LG, Lai WW, Afilalo J, Hua L, Handschumacher MD, Chandrasekaran K, Solomon SD, Louie EK, Schiller NB. Guidelines for the echocardiographic assessment of the right heart in adults: a report from the American Society of Echocardiography endorsed by the European Association of Echocardiography, a registered branch of the European Society of Cardiology, and the Canadian Society of Echocardiography. J Am Soc Echocardiogr. 2010 Jul;23(7):685-713; quiz 786-8. doi: 10.1016/j.echo.2010.05.010. No abstract available. PMID 20620859
- [Background] St-Pierre P, Deschamps A, Cartier R, Basmadjian AJ, Denault AY. Inhaled milrinone and epoprostenol in a patient with severe pulmonary hypertension, right ventricular failure, and reduced baseline brain saturation value from a left atrial myxoma. J Cardiothorac Vasc Anesth. 2014 Jun;28(3):723-9. doi: 10.1053/j.jvca.2012.10.017. Epub 2013 Apr 26. No abstract available. PMID 23623891